CLINICAL TRIAL: NCT06484842
Title: A Randomised Controlled Study to Evaluate the Effectiveness of the Combined Psychological Resilience and Self-efficacy Intervention for Oesophageal Cancer Surgery Patients
Brief Title: Evaluation of the Effectiveness of the Combined Psychological Resilience and Self-efficacy Intervention for Improving Resilience and Self-efficacy and Reducing Anxiety and Depression of Oesophageal Cancer Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Collaborators: Anhui Medical University School of Nursing Qingmiao Programme (Unknown); Natural Science Foundation of Anhui Provincial Department of Education (Unknown)
Responsible Party: Principal Investigator, Jinghan Zhao, Master candidate, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 83242327
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Neoplasms; Resilience, Psychological; Self Efficacy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The combined intervention group (Experimental): The combined intervention group will receive the combined psychological resilience and self-efficacy intervention.
  Interventions: Other: The combined psychological resilience and self-efficacy intervention
- The single intervention group (Experimental): The single intervention group will receive the mindfulness intervention.
  Interventions: Other: The mindfulness intervention
- The control group (No Intervention): The control group will receive routine care. Routine care mainly includes postoperative precautions, management of postoperative complications, and postoperative dietary care such as the type, time, and amount of food required, etc. In addition, we will add the patients' WeChat and send relevant health knowledge to the patients regularly. The control group theoretically will not receive any additional psychological interventions. However, they will be entitled to receive either the combined psychological resilience and self-efficacy intervention or the psychological resilience intervention once the combined and single intervention groups have completed the intervention.

INTERVENTIONS:
Other: The combined psychological resilience and self-efficacy intervention — Based on the content of the literature analysis and the group's previous research, a joint intervention programme on psychological resilience and self-efficacy for patients undergoing surgery for oesophageal cancer has been developed. The programme consists of 6 sessions in total, including preoperative period and one month after discharge, covering the period when patients' postoperative symptoms occur most severely. The intervention will be conducted in an individual, offline face-to-face format during the patients' hospital stay; considering the smooth implementation of the intervention after the patient will be discharged from the hospital, we will conduct the intervention in an individual, offline face-to-face format during the patient's outpatient review, and set up a WeChat group in case the patients are at home to conduct the intervention in the form of an online punch card.
  Arms: The combined intervention group
Other: The mindfulness intervention — The oesophageal cancer surgery patients in the single intervention group will receive 5 sessions of mindfulness intervention consistent with the mindfulness intervention component of the combined intervention programme. The intervention will be conducted in an individual, offline face-to-face format during the patients' hospitalisation; we will conduct the intervention in an individual, offline face-to-face format during the patients' outpatient review, and set up a WeChat group in case the patients are at home in the form of an online punch card. Each session will include a pre-session reflection and post-session homework. The whole process will be supervised and reminded by interventionists, who will respond to patients' questions in a timely manner to ensure patients safety and the smooth implementation of the intervention. Adjustments and improvements will be made at any time according to the needs of patients undergoing oesophageal cancer surgery.
  Arms: The single intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the combined psychological resilience and self-efficacy intervention in oesophageal cancer surgery patients. The main question it aims to answer is:

Is the combined psychological resilience and self-efficacy intervention program more effective than the single psychological resilience intervention in improving psychological resilience and self-efficacy and reducing anxiety and depression in patients undergoing oesophageal cancer surgery? Researchers will compare the combined psychological resilience and self-efficacy intervention program to the single psychological resilience intervention and routine care to see if the combined intervention can improve psychological resilience and self-efficacy and reduce anxiety and depression in oesophageal cancer surgery patients.

Participants will receive the combined psychological resilience and self-efficacy intervention program in the combined intervention group, the single psychological resilience intervention in the single intervention group and routine care in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with oesophageal cancer by pathological biopsy.
* Received surgical treatment.
* Native Chinese speakers and age≥18 years old.

Exclusion Criteria:

* Prior to or during the first evaluation, patients who had end-stage illnesses or other chronic ailments including kidney failure, heart failure, etc..
* Undergoing further supplementary therapies such as neoadjuvant chemotherapy or radiotherapy.
* Undergoing other systematic psychological therapies.
* Possess a background of psychopathy or cognitive problems.
* Patients' baseline anxiety and depression subscale scores are less than 8 points each.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Psychological resilience | before the intervention (T0: 1-3 days before surgery), during the intervention (T1: 7 days after surgery), and after the intervention (T2: 2-3 weeks after discharge)
  Psychological resilience will be measured using the Connor-Davidson Resilience Scale (CD-RISC), which was developed by American psychologists Connor and Davidson in 2003 based on a research project on post-traumatic stress disorder to measure the level of psychological resilience in the general population and in clinical patients over the past month. It is now widely used to measure levels of psychological resilience in patients with cancer and chronic diseases. The scale consists of 25 items, including three dimensions of resilience, self-improvement, and optimism, and each item is scored on a 5-point Likert scale, with scores of 0-4 indicating from "not true at all" to "true nearly all the time". The total score ranges from 0 to 100, and the higher the score, the higher the psychological resilience. In 2007, Yu Xiaonan and other scholars translated it into Chinese, and the Cronbach's α coefficient was 0.91.
Self-efficacy | before the intervention (T0: 1-3 days before surgery), during the intervention (T1: 7 days after surgery), and after the intervention (T2: 2-3 weeks after discharge)
  Self-efficacy will be measured using the General Self-Efficacy Scale (GSES), which was first developed in 1981 by Professor Schwarzer, a leading clinical and health psychologist at the Freie Universität Berlin, Germany, and his colleagues, and has now been translated into several languages and adopted worldwide. At first, it consisted of 20 items with a 4-point scale, but later it was improved to 10 items with a Likert scale of 1-4, ranging from "not at all true" to "exactly true", with higher overall scores indicating stronger self-efficacy of the individual. The scale was translated into Chinese by our scholars Zhang Jianxin and Schwarzer in 1995, and Chineseised by a Chinese scholar Wang Caikang in 2001, with a total of 10 items, an internal consistency coefficient of 0.87, a re-test reliability of 0.83 at an interval of about 10 days, and a half-way reliability of 0.90.

SECONDARY OUTCOMES:
Anxiety and depression | before the intervention (T0: 1-3 days before surgery), during the intervention (T1: 7 days after surgery), and after the intervention (T2: 2-3 weeks after discharge)
  Anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS), which was developed by Zigmond et al. in 1983 and is a simple and easy-to-use scale with good reliability, validity, and psychometric properties. It consists of two subscales, anxiety and depression, with a total of 14 entries, of which 7 entries (single number) assess anxiety and 7 entries (double number) assess depression, and it is a self-assessment 4-rating scale, i.e., each entry is divided into four rating scales, which are recorded as 0, 1, 2, and 3, respectively, and the total scores of both anxiety and depression subscales range from 0-21. This scale was introduced to China in 1993 by Ye Weifei and other scholars, and was revised and translated into a Chinese version suitable for the Chinese population, with reliability analyses confirming that the coefficients of the anxiety and depression subscales were 0.72 and 0.68, and the total Cronbach's α coefficient was 0.785.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06484842/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT06484842/ICF_001.pdf